CLINICAL TRIAL: NCT06028919
Title: A Randomised Control Trial of Power Versus Temperature-controlled Irrigated Radiofrequency Ablation for the Treatment of Ventricular Tachycardia (VT)
Brief Title: Power Versus Temperature Controlled Ablation for Treatment of VT
Acronym: DTinVT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Medtronic (Industry); Coventry University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TS584122
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ventricular Tachycardia
Keywords: temperature controlled irrigated radiofrequency ablation; ventricular tachycardia; clinical outcomes
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: patient-blinded, prospective, multi centre, two-arm, randomised controlled trial
Who Masked: Participant
Masking Description: The patient will be blinded to which trial arm they have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Temperature controlled DiamondTemp (DT) ablation catheter (Other): Intervention arm
  Interventions: Device: Temperature controlled DiamondTemp (DT) ablation catheter
- Power controlled Tacticath/Tactiflex ablation catheter (Other): Control arm
  Interventions: Device: Tacticath/Tactiflex (TF) ablation catheter

INTERVENTIONS:
Device: Temperature controlled DiamondTemp (DT) ablation catheter — The DiamondTemp catheter is a new ablation catheter that uses 6 industrial grade diamonds to actually measure the temperature of the surface tissue being cauterised. This enables the DiamondTemp catheter to control the amount of power being delivered from the ablation catheter into the tissue being ablated by maintaining a constant temperature at the surface of the heart.
  Arms: Temperature controlled DiamondTemp (DT) ablation catheter
Device: Tacticath/Tactiflex (TF) ablation catheter — The Tactiflex ablation catheter is currently the market leader and routinely used for VT ablation.
  Arms: Power controlled Tacticath/Tactiflex ablation catheter

SUMMARY:
Ventricular Tachycardia (VT) is a life threatening heart rhythm that comes from the bottom chambers of the heart (the ventricles) and is a leading cause of sudden cardiac death.

The majority of patients that are at risk of VT or suffer a cardiac arrest will have an Internal Cardiac Defibrillator (ICD) in situ to treat the abnormal heart rhythm. The ICD can deliver a painful shock to restore normal heart rhythm but importantly does not treat the underlying cause. Current treatment for the prevention of recurrent VT include catheter ablation (CA) or medication. Long-term results with global 12 month VT-free survival rates with CA are around 50%.

The trial is to compare 2 different types of ablation catheter that are used to cauterise small areas of unhealthy tissue within the heart that are responsible for VT: Diamond Temp (DT) and Tacticath/Tactiflex (TF). Our hypothesis is that the DT ablation catheter will provide comparable efficacy and safety for the treatment of VT as the current industry gold standard (TF).

DETAILED DESCRIPTION:
This trial compares 2 different types of ablation catheter for the treatment of ventricular tachycardia (VT). VT is a life threatening heart rhythm that comes from the bottom chambers of the heart (the ventricles) and is associated with poor patient prognosis, outcomes and is a leading cause of sudden cardiac death in developed countries.

Current treatments for VT include catheter ablation (CA), medication and having an internal cardiac defibrillator (ICD) implanted, each treatment has advantages and disadvantages. The ICD can deliver a lifesaving shock but this doesn't treat the cause of the VT and can be very painful and upsetting for the patient. Medications can reduce the amount and rate of VT but can have dangerous side effects.

CA involves small tubes being placed in the heart and small areas of unhealthy heart tissue are burnt (ablated) to stop the VT. This is the only treatment that treats the underlying cause but long-term success is about 50% after 1 year.

The investigators want to improve the success rates of VT ablation. There is a new ablation catheter called Diamond Temp which works differently to the current industry gold standard (Tacticath/Tactiflex Catheter). The investigators think the Diamond Temp catheter will be better than the Tacticath catheter but need to do this trial to prove it.

This trial will be at University Hospital Coventry and Warwickshire and University Hospitals Sussex involving patients that suffer VT, have an ICD and need an ablation. If a patient wishes to participate they will give consent and be chosen at random to receive ablation with either Diamond temp or Tacticath/Tactiflex. All other treatment will be the same as after a normal ablation procedure. Participants will be followed up at 6 months and 1 year after the procedure as well as being monitored by the ICD clinic. The study will have 54 patients and be completed in 2025.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age to give informed consent specific to national legal requirements.
* Subject with 1 of the following:

  1. Symptomatic VT (despite optimal medical therapy), 3 or more episodes of VT within 24 h (VT storm).
  2. At least 3 episodes of VT requiring anti-tachycardia pacing (ATP)
  3. At least one appropriate ICD shock.
* Referred for VT ablation by Consultant Electrophysiologist
* Subject discussed at cardiac EP MDT
* Suitable candidate for intra-cardiac mapping and ablation of arrhythmia.
* Subject agrees to comply with study procedures and be available for routine follow up visits for at least 12 months after enrolment.
* Subject is willing and able to provide written consent

Exclusion Criteria:

* BMI >40kg/m2
* Presence of intramural thrombus, tumour or abnormality that precludes vascular access, catheter introduction or manipulations.
* Coagulopathy, bleeding diathesis or suspected pro-coagulant state.
* Sepsis, active systemic infection or fever (>100.5 F/38 C) within a week prior to the ablation procedure.
* Significant restrictive or obstructive pulmonary disease or chronic respiratory condition.
* Renal failure requiring dialysis or renal compromise that in the investigators judgement would increase risk to the subject or deem the subject inappropriate to participate in the study.
* Known allergies or intolerance to anticoagulant and antiplatelet therapies to be used in conjunction with the study or contrast sensitivity that can't be adequately pre-treated prior to the ablation procedure.
* Positive pregnancy test results for female subjects of childbearing or potential or breast feeding.
* Enrolment in a concurrent clinical study that in the judgement of the investigator would increase risk to the subject or deem the subject inappropriate to participate in the study.
* Significant GI bleed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the efficacy of the DT versus the TF ablation catheter for the treatment of VT | 12 months post ablation
  The efficacy of each ablation catheter will be compared by measuring the VT burden 12 months post-ablation.
Assessing the safety of the DT versus the TF ablation catheter for the treatment of VT | within 30 days or 6 months after index ablation procedure
  The efficacy of each ablation catheter will be compared by measuring the freedom from a composite of pre-specified procedure-related complications (adverse outcomes).

SECONDARY OUTCOMES:
Perceived health benefit of treatment | at baseline and 12 months
  The patient's health benefit will be measured using a EQ-5D-5L questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Tarv Dhanjal, PhD, Principal Investigator — University Hospitals Coventry and Warwickshire NHS Trust
Locations (2):
- United Kingdom (2):
  - University Hospital Coventry and Warwickshire NHS Trust, Coventry, West Midlands
  - University Hospitals Sussex NHS Foundation Trust, Brighton

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.